CLINICAL TRIAL: NCT00601705
Title: A Phase II Trial of Induction Chemotherapy With Epirubicin, Oxaliplatin and Fluorouracil (EOF) Followed by Esophagogastrectomy and Post-operative Concurrent Chemoradiotherapy With Fluorouracil and Cisplatin, in Patients With Loco-regionally Advanced Adenocarcinoma of the Esophagus, Gastroesophageal Junction and Gastric Cardia
Brief Title: Epirubicin, Oxaliplatin and Fluorouracil (EOF) in Cancer of the Esophagus, Gastroesophageal Junction, or Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2Y07; P30CA043703 (NIH); CASE2Y07 (Other: Case Comprehensive Cancer Center); NCI-2010-01196 (Other: NCI/CTRP)
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: adenocarcinoma of the esophagus; adenocarcinoma of the stomach; stage III esophageal cancer; stage IV esophageal cancer; stage III gastric cancer; stage IV gastric cancer; stage II esophageal cancer; stage II gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Epirubicin; Fluorouracil; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epirubicin, Oxaliplatin and Fluorouracil (Experimental)
  Interventions: Drug: cisplatin; Drug: epirubicin hydrochloride; Drug: fluorouracil; Drug: oxaliplatin; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy

INTERVENTIONS:
Drug: cisplatin — 20 mg/m2/day IV continuous infusion over 24 hours for 96 total hours.
Drug: epirubicin hydrochloride — 50 mg/m2 IV bolus
Drug: fluorouracil — 200 mg/m2/day will be given as a continuous intravenous infusion for all 9 weeks, beginning on day 1.
Drug: oxaliplatin — 130 mg/m2 IV infusion over 2 hours
Procedure: adjuvant therapy — Between 6-10 weeks after surgery patients will begin postoperative chemoradiotherapy. Daily radiation therapy fractions of 180-200 cGy will be given to the esophago-gastric bed and draining lymphatic regions to a total dose of 50-55 Gy (60 Gy in the event of an R1 or R2 resection). Concurrent with this radiation, two cycles of chemotherapy will be given, during the first and fourth weeks of the radiation
Procedure: neoadjuvant therapy — Three weeks after discontinuing the fluorouracil (12 weeks after study entry) patients will be fully restaged to assess for a clinical response, and to ensure that there is no contraindication to surgical resection, which will be scheduled for approximately one week later (13 weeks after study entry).
  Surgery will consist of a transthoracic esophagogastrectomy or a total gastrectomy with Roux-en-Y esophagojejunostomy depending on the location and extent of the tumor at surgery. An appropriate lymphadenectomy will be performed. Immediate reconstruction is anticipated if possible.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin, oxaliplatin, fluorouracil, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy and radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy, surgery, and radiation therapy works in treating patients with locoregionally advanced cancer of the esophagus, gastroesophageal junction, or stomach.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility and tolerability of induction chemotherapy comprising epirubicin hydrochloride, oxaliplatin, and fluorouracil (EOF), followed by surgical resection and postoperative concurrent chemoradiotherapy comprising fluorouracil and cisplatin in patients with locoregionally advanced adenocarcinoma of the esophagus, gastroesophageal junction, or gastric cardia.

Secondary

* To determine the rate of complete and partial response to three courses of EOF induction chemotherapy.
* To compare the recurrence-free and overall survival of patients treated with this regimen vs historical controls at this institution.
* To compare patterns of failure in patients treated with this regimen vs historical controls at this institution.

OUTLINE:

* Induction chemotherapy: Patients receive epirubicin hydrochloride IV over 3-15 minutes and oxaliplatin IV over 2 hours on day 1 and fluorouracil IV continuously on days 1-21. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
* Surgery: Four weeks after completion of induction chemotherapy, patients with locoregionally confined disease (T0-4, N0-1, M0-1a) undergo transthoracic esophagogastrectomy or total gastrectomy with Roux-en-Y esophagojejunostomy, depending on the location and extent of the tumor at the time of surgery.
* Postoperative chemoradiotherapy: Beginning 6-10 weeks after surgery, patients undergo radiotherapy 5 days a week for approximately 6 weeks. Patients also receive fluorouracil IV continuously and cisplatin IV continuously over 96 hours in weeks 1 and 4 of radiotherapy.

After completion of study treatment, patients are followed every 8-12 weeks for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologic diagnosis of adenocarcinoma of the esophagus, gastroesophageal junction or gastric cardia, based on biopsy material or adequate cytologic exam.
* Patients must be clinically staged according to the AJCC 2002 staging system and must have either T3-4, or N1 or M1a disease. Staging should include at least an upper endoscopy with endoscopic ultrasound and an FDG-PET/CT scan.
* Patients must have an ECOG performance status of 0-1.
* Patients must have adequate bone marrow function as evidenced by: Absolute neutrophil count > 1,500/uL Platelet count > 100,000/uL
* Patients must have adequate renal function as evidenced by serum creatinine < 1.6 mg/dL
* Patients must have adequate hepatic function as evidenced by:Serum total bilirubin < 1.5 mg/dL Alkaline phosphatase < 3X the institutional ULN AST/ALT < 3X the institutional ULN
* Patients must have adequate pulmonary function as evidenced by an FEV1 > 50% predicted.
* Patients or their legal representatives must be able to read, understand, provide and sign informed consent to participate in the trial.
* Patients of childbearing potential agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method)
* Age > 18 years

Exclusion Criteria:

* Patients with any other diagnosis except for adenocarcinoma (squamous cell carcinoma, small cell carcinoma, mixed adenosquamous, lymphoma, sarcoma etc,) will be ineligible.
* Patients with any evidence of distant hematogenous or distant nodal disease (M1b) will be ineligible.
* No prior chemotherapy, radiation therapy or surgery for this malignancy will be allowed. Prior endoscopic debulking, laser therapy or dilatation will not exclude a patient.
* Patients with another active malignancy will not be eligible except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current PSA of < 1.0 mg/dL on 2 successive evaluations at least 3 months apart, with the most recent evaluation within 4 weeks of entry
* Patients with an active infection will not be eligible.
* Patients with known hypersensitivity to any of the components of oxaliplatin, epirubicin, fluorouracil or cisplatin will not be eligible.
* Patients who are receiving any other concurrent investigational therapy, or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication) will not be eligible.
* Patients with a baseline peripheral neuropathy greater than or equal Grade 2 will not be eligible.
* Patients who are pregnant or lactating will not be eligible.
* Patients with any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results, will not be eligible.
* Patients with any history of an allogeneic transplant will not be eligible.
* Patients with known infection with HIV, Hepatitis B or C (active, previously treated or both) will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-01-05 (Actual); Primary Completion 2012-03-26 (Actual); Study Completion 2015-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Adelstein, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Epirubicin, Oxaliplatin, 5-fluorouracil, and Surgery: Subjects received epirubicin (50-mg/m^2), oxaliplatin (130-mg/m^2), 5-fluorouracil (5FU; 200mg/m^2/d), and surgery, which took place 4 to 5 weeks after the completion of preoperative chemotherapy. Epirubicin and oxaliplatin were given on day 1, while 5FU was intravenously infused for 21-days. Surgery was conducted 4 to 5-weeks after chemotherapy. Six to ten-weeks after surgery chemoradiotherapy was initiated. With radiotherapy, patients received two cycles of cisplatin and 5FU during the first and fourth weeks after surgery; they were administered intravenously over 96-hours. Specifically, cisplatin and 5FU total dose was 80-mg/m^2 (20-mg/m^2/d) and 4000 mg/m^2 (1000-mg/m^2/d), respectively.
Period: Overall Study
Arm/Group | Epirubicin, Oxaliplatin, 5-fluorouracil, and Surgery
Started | 61
Completed | 60
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Epirubicin, Oxaliplatin, 5-fluorouracil, and Surgery
Number analyzed (Participants) | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [37 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Induction Chemoradiotherapy as Measured by Resectability Rate
Description: Feasibility of induction chemoradiotherapy as measured by resectability in greater than 75% of participants. The number of participants that were resectable.
Time Frame: at 12 weeks from on study
Population: All subjects that went on study and received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Epirubicin, Oxaliplatin, 5-fluorouracil, and Surgery
Number analyzed (Participants) | 60
Participants | 54

2. Secondary Outcome: Clinical Response Rate
Description: Percent of participants with a clinical response:
  Complete clinical response is defined as the complete disappearance of all clinical evidence of tumor.
  Partial clinical response is defined as any improvement in the clinically determined T or N stage (without reciprocal deterioration in N or T) or a resolution of M1a disease, when compared to the pretreatment clinical stage. A partial response will not be defined based only on shrinkage of a measurable lesion unless there is improvement in the TNM stage.
  Stable clinical disease is defined as no change in the clinical TNM stage when compared to the pretreatment clinical stage.
  Progressive clinical disease is defined as any increase in the T or N stage irrespective of any reciprocal improvement in N or T, or as the development of new areas of malignancy or metastases.
Time Frame: at 12 weeks from on study
Population: Participants that complete induction therapy
Measure: Number; unit: percentage of participants
Groups:
- Epirubicin, Oxaliplatin and Fluorouracil: Epirubicin, Oxaliplatin and Fluorouracil (EOF) followed by Esophagogastrectomy and post-operative concurrent chemoradiotherapy with Fluorouracil and Cisplatin
Arm/Group | Epirubicin, Oxaliplatin and Fluorouracil
Number analyzed (Participants) | 58
percentage of participants
  Complete response | 0
  Partial response | 48
  Stable disease | 33
  Progressive disease | 19

3. Secondary Outcome: Pathological Response Rate
Description: Percent of participants with a clinical response:
  Complete pathologic response is defined as the complete disappearance of all viable tumor in the surgical specimen.
  Partial pathologic response is defined as any improvement in the pathologically determined T or N stage (without reciprocal deterioration in N or T) or a resolution of M1a disease, when compared to the pretreatment esophageal ultrasound-determined clinical stage. A partial response will not be defined based only on shrinkage of a measurable lesion unless there is improvement in the TNM stage.
  Stable pathologic disease is defined as no change in the pathologically determined TNM stage when compared to the pretreatment esophageal ultrasound.
  Progressive pathologic disease is defined as any increase in the T or N stage irrespective of any reciprocal improvement in N or T, or as the development of new areas of malignancy or metastases.
Time Frame: after completion of study at 35 weeks
Population: Participants that complete induction therapy
Measure: Number; unit: participants
Arm/Group | Epirubicin, Oxaliplatin and Fluorouracil
Number analyzed (Participants) | 58
participants
  Complete response | 3
  Partial response | 21
  Stable disease | 14
  Progressive disease | 20

4. Secondary Outcome: Overall Survival
Description: Percent of participants with a 3-year survival. A survival rate greater than 50% would suggest efficacy and justify further study.
Time Frame: at 3 years from on study
Population: All patients that went on study
Measure: Number; unit: percentage of participants
Arm/Group | Epirubicin, Oxaliplatin, 5-fluorouracil, and Surgery
Number analyzed (Participants) | 60
percentage of participants | 47

5. Secondary Outcome: Locoregional Control and Distant Metastatic Control
Description: A distant metastatic control rate of greater than 55 % would suggest efficacy for this treatment protocol. A locoregional control rate of less than 75% would suggest inefficacy. Locoregional control (LRC) defined by recurrence at the primary site or in regional lymph nodes and distant metastatic control (DMC), defined by recurrence in a distant site.
Time Frame: at 3 years from on study
Population: All participants that went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Epirubicin, Oxaliplatin, 5-fluorouracil, and Surgery
Number analyzed (Participants) | 60
Participants
  Locoregional Control | 4
  Distant Metastatic Control | 29

6. Secondary Outcome: Postoperative Adjuvant Chemoradiotherapy Feasibility
Description: Ability to complete postoperative chemoradiotherapy. A threshold level of 65% was set and if less than this percentage completed the phase, it would be deemed unacceptable. The anticipation was that 53-patients would be evaluable for this end point.
Time Frame: Between 6 to 10 weeks postoperatively
Population: All patients that went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Epirubicin, Oxaliplatin, 5-fluorouracil, and Surgery
Number analyzed (Participants) | 60
Participants | 48

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events while on study, treatment and the 30 days following treatment discontinuation over a period of up to 1 year.
Description: Adverse events were reported separately for pre-operative therapy (60 participants) and post-operative therapy (48 participants).
Groups:
- Epirubicin, Oxaliplatin and Fluorouracil: cisplatin: 20 mg/m2/day IV continuous infusion over 24 hours for 96 hours.
  epirubicin hydrochloride: 50 mg/m2 IV bolus
  fluorouracil: 200 mg/m2/day continuous infusion for all 9 weeks, beginning on day 1.
  oxaliplatin: 130 mg/m2 IV infusion over 2 hours
  adjuvant therapy: At 6-10 weeks after surgery patients will begin postoperative chemoradiotherapy. Daily radiation therapy fractions of 180-200 cGy will be given. Concurrent with this radiation, two cycles of chemotherapy will be given, during the first and fourth weeks of the radiation
  neoadjuvant therapy: Three weeks after discontinuing the fluorouracil patients will be fully restaged to assess for a clinical response, and to ensure that there is no contraindication to surgical resection, which will be scheduled for app
Arm/Group | Epirubicin, Oxaliplatin and Fluorouracil
All-Cause Mortality (participants affected / at risk) | 41/60
Serious Adverse Events (participants affected / at risk) | 24/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epirubicin, Oxaliplatin and Fluorouracil (N=60)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (11)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Enteritis - inflammation of the small bowel (Gastrointestinal disorders) | 2 (2)
Fistula, GI - Stomach (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis - oral cavity (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (9)
Vomiting (Gastrointestinal disorders) | 4 (9)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Colitis, infectious (Infections and infestations) | 1 (1) — Clostridium Difficile
Neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) — fainting
Thrombosis (Vascular disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Epirubicin, Oxaliplatin and Fluorouracil (N=60)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 8/48 — Postoperative therapy
pneumonia (Respiratory, thoracic and mediastinal disorders) | 8/48 — Postoperative therapy
wound infections (Injury, poisoning and procedural complications) | 10/48 — Postoperative therapy
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 9 — Preoperative therapy
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 9/48 — Postoperative therapy
Neutropenia (Blood and lymphatic system disorders) | 19 — Preoperative therapy
Neutropenia (Blood and lymphatic system disorders) | 13/48 — Postoperative therapy
Febrile neutropenia (Blood and lymphatic system disorders) | 5/48 — Postoperative therapy
Platelets <50,000/μl (Blood and lymphatic system disorders) | 10/48 — Postoperative therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes